CLINICAL TRIAL: NCT02210052
Title: Safety of Lumbar Spine Radiofrequency Procedures in the Presence of Posterior Pedicle Screws: A Prospective Trial
Brief Title: Safety of Spine Radiofrequency Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tim J. Lamer, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14-003619
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Radiofrequency Ablation in Patients With Spinal Hardware
Keywords: radiofrequency ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiofrequency neurotomy subjects (Experimental): Subjects with spinal hardware that are undergoing radiofrequency ablation procedures will have an additional radiofrequency cannula placed at the site of adjacent pedicle screws for temperature measurement only.
  Interventions: Device: Radiofrequency cannula

INTERVENTIONS:
Device: Radiofrequency cannula — Subjects with spinal hardware that are undergoing radiofrequency ablation procedures will have an additional radiofrequency cannula placed at the site of adjacent pedicle screws for temperature measurement only.

SUMMARY:
The goal of the study was to determine if patients undergoing radiofrequency neurotomy (RFN) of lumbar facet joints that are adjacent to previously placed pedicle screws from a fusion, would lead to an increase in the temperature of the pedicle screws.

DETAILED DESCRIPTION:
This study was a prospective clinical trial, examining outcomes related to temperature increases in pedicle screws. It was not possible to blind the investigators or the patient. Outcomes related temperature differences were collected at each pedicle screw adjacent to a zygapophyseal joint being treated.

A conventional 18-gauge, 1-cm curved active tip radiofrequency cannula was placed under fluoroscopic guidance to the area to be treated (the junction of the transverse process and the superior articulating process of the facet joint). This position placed the tip of the radiofrequency cannula immediately adjacent to, but not in direct contact with, the pedicle screws. The radiofrequency cannula was connected to a radiofrequency generator, and the conventional settings for clinical medial branch neurotomy was used, heating the tissue to 80°C for 90 seconds. The procedure described up to this point is the normal procedure and protocol for RFN performed at the Mayo Clinic.

The experimental portion of the procedure is as follows: A separate 22 gauge radiofrequency cannula was intentionally placed in direct contact with the dorsal surface of the pedicle screws and was connected to a radiofrequency generator solely for the purpose of measuring temperature, as the RF cannula are dual purpose probes capable of both conducting energy for the radiofrequency lesion and monitoring tissue temperature. In other words, this small gauge needle was placed for the sole purpose of acting as a thermistor probe/temperature monitor. This process was repeated for each level necessary for treatment.

ELIGIBILITY:
Inclusion Criteria:

- Scheduled for Radiofrequency procedure AND has spinal hardware placed from a previous spinal surgery

Exclusion Criteria:

* Active infection over skin where needle will be placed
* Coagulopathy
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim J Lamer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gazelka HM, Welch TL, Nassr A, Lamer TJ. Safety of lumbar spine radiofrequency procedures in the presence of posterior pedicle screws: technical report of a cadaver study. Pain Med. 2015 May;16(5):877-80. doi: 10.1111/pme.12678. Epub 2015 Jan 8. PMID 25580992
- [Result] Lamer TJ, Smith J, Hoelzer BC, Mauck WD, Qu W, Gazelka HM. Safety of Lumbar Spine Radiofrequency Procedures in Patients Who Have Posterior Spinal Hardware. Pain Med. 2016 Sep;17(9):1634-7. doi: 10.1093/pm/pnv078. Epub 2016 Jan 13. PMID 26764338

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiofrequency Neurotomy Subjects
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiofrequency Neurotomy Subjects
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 47.8 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Procedures in Which Temperature of Screws Increased
Description: The study will measure for increased temperature in pedicle screws adjacent to lumbar facet joints during radiofrequency neurotomy (RFN). Temperatures will be recorded by placing a thermistor probe on the surface of the adjacent hardware.
Time Frame: 2 hours
Population: There were 6 participants, but some participants had more than 1 procedure. There were a total of 10 procedures analyzed.
Measure: Number; unit: procedures
Units Other Than Participants: Procedures
Arm/Group | Radiofrequency Neurotomy Subjects
Number analyzed (Participants) | 6
Number analyzed (Procedures) | 10
procedures
  Non-significant increase | 4
  Significant increase; procedure stopped | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collect during the procedure.
Arm/Group | Radiofrequency Neurotomy Subjects
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes